CLINICAL TRIAL: NCT00814736
Title: A Randomized, Double-Blinded, Placebo-Controlled, Two-Way Crossover Study to Investigate The Safety And Toleration Of Single Dose Sildenafil In Subjects Receiving Chronic UK-369,003.
Brief Title: A Randomized, Double-Blinded, Placebo-Controlled, Two-Way Crossover Study to Investigate the Safety and Toleration of Single Dose Sildenafil in Subjects Receiving Chronic UK-369,0031
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: A3711051
Record Dates: First submitted 2008-11-03; First posted 2008-12-25 (Estimated); Last update posted 2008-12-25 (Estimated); Status verified 2008-12

CONDITIONS: Prostatic Hyperplasia; Urinary Bladder, Overactive; Erectile Dysfunction
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder, Overactive; Erectile Dysfunction | interventions — 1-(6-ethoxy-5-(3-ethyl-6,7-dihydro-2-(2-methoxyethyl)-7-oxo-2H-pyrazolo(4,3-d)pyrimidin-5-yl)-3-pyridyl sulphonyl)-4-ethylpiperazine; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- UK369,003 + Placebo or sildenafil (Experimental): All subjects will receive 17 days daily dosing of UK-369,003 100 mg MR Subjects will receive single oral doses of the following interactant treatments in a randomized order On Day 14, a single dose of sildenafil-matching placebo or 100 mg sildenafil and on Day 17 a single dose of 100 mg sildenafil or a sildenafil matching placebo
  Interventions: Drug: UK369,003; Drug: sildenafil; Drug: sildenafil matching placebo

INTERVENTIONS:
Drug: UK369,003 — oral tablet, once a day
Drug: sildenafil — single oral dose on day 14 or day 17
  Other Names: viagra
Drug: sildenafil matching placebo — single oral dose on day 14 or day 17

SUMMARY:
To investigate the safety and overall tolerability of co-administration two PDE5 inhibitors UK369,003 and sildenafil

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Healthy male subjects between the ages of 40 and 55 years, inclusive
* Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Loss of vision in one eye due to non-arteritic ischemic optic neuropathy (NAION) regardless of whether or not this event was temporally associated with the use of a PDE5 inhibitor.

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety and toleration assessed by non-leading questioning, incidence of adverse events and laboratory testing. | hours

SECONDARY OUTCOMES:
Incidence of postural hypotension. | hours
Standing and supine pulse rate (PR) at each postdose time. | hours
Standing systolic and diastolic blood pressure (BP) and supine systolic and diastolic BP at each postdose time. | hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3711051&StudyName=A%20randomized%2C%20double-blinded%2C%20placebo-controlled%2C%20two-way%20crossover%20study%20to%20investigate%20the%20safety%20and%20toleration%20of%20single%20dose%20Silden